CLINICAL TRIAL: NCT02743130
Title: Postprandial Glycemic Response to Berry Nectars Containing Inverted Sugar
Brief Title: Effects of Berry Nectars Sweetened With Inverted Sugar on Post-meal Blood Sugar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Finnsugar Ltd (Unknown)
Responsible Party: Principal Investigator, Riitta Törrönen, Senior Scientist, University of Eastern Finland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: INVE 903/020502/2014
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Hyperglycemia, Postprandial
Keywords: Berries; Blackcurrant (Ribes nigrum); Lingonberry (Vaccinium vitis-idaea); Sucrose; Inverted sugar; Postprandial glucose response; Postprandial insulin response
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blackcurrant nectar (Experimental): Contains 17.5 g glucose and 17.5 g fructose representing 35 g completely inverted sucrose
  Interventions: Dietary Supplement: Blackcurrant Nectar
- Lingonberry nectar (Experimental): Contains 17.5 g glucose and 17.5 g fructose representing 35 g completely inverted sucrose
  Interventions: Dietary Supplement: Lingonberry Nectar
- Reference (Active Comparator): Sugar control, contains 17.5 g glucose and 17.5 g fructose in water
  Interventions: Dietary Supplement: Reference

INTERVENTIONS:
Dietary Supplement: Blackcurrant Nectar — Consumption of a single dose (300 ml)
  Arms: Blackcurrant nectar
Dietary Supplement: Lingonberry Nectar — Consumption of a single dose (300 ml)
  Arms: Lingonberry nectar
Dietary Supplement: Reference — Consumption of a single dose (300 ml)
  Arms: Reference

SUMMARY:
Berries have been shown to improve postprandial glucose and insulin responses to sucrose. During processing and storage of berry products, sucrose is inverted to glucose and fructose. The effects of berries on the glycemic response induced by inverted sugar are not known. The purpose of this study is to determine whether berries are effective in lowering the postprandial glucose and insulin responses induced by inverted sugar.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-28 kg/m2
* Normal fasting plasma glucose

Exclusion Criteria:

* Smoking
* Diabetes or other chronic disease
* Antibiotic medication within the past 3 months
* Blood donation within the past month

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Plasma glucose response | 2 hours
  0, 15, 30, 45, 60, 90, 120 minutes post-meal

SECONDARY OUTCOMES:
Plasma insulin response | 2 hours
  0, 15, 30, 45, 60, 90, 120 minutes post-meal

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Törrönen, Dr, Principal Investigator — Senior Scientist
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No